CLINICAL TRIAL: NCT00331474
Title: The Effect of BCG Vaccination on Immune Responses in HIV-Exposed and Unexposed Infants
Brief Title: The Effect of Bacille Calmette Guerin (BCG) Vaccination on Immune Responses in HIV-Exposed and Unexposed Infants
Status: Unknown | Phase: Phase 1 / Phase 2 | Type: Interventional
Last Known Status: Active, not recruiting
Sponsor: University of Stellenbosch (Other)
Collaborators: Thrasher Research Fund (Other)
Responsible Party: Esther Steyn or Liesel Strauss, Stellenbosch University
Allocation: Randomized | Model: Parallel | Masking: None | Purpose: Prevention
Other Study IDs: N06/04/071
Record Dates: First submitted 2006-05-30; First posted 2006-05-31 (Estimated); Last update posted 2009-02-16 (Estimated); Status verified 2009-02

CONDITIONS: HIV Infections
Keywords: BCG; HIV; Immune responses; Delayed vaccination; Infant morbidity; Nutritional status; Morbidity; Mortality
MeSH Terms: conditions — HIV Infections

INTERVENTIONS:
Biological: BCG delayed — early (birth) and delayed (14 weeks) intradermal BCG vaccination
  Other Names: early vs. delayed BCG

SUMMARY:
Background:

Each year, more than half a million babies are infected with HIV by mother-to child transmission in developing countries. Many of these babies get sick and develop HIV disease (AIDS) at a very young age. Exposure to other infectious diseases may influence this early progression to AIDS. BCG is a live tuberculosis vaccine made from cow tuberculosis. It is routinely given at birth to most babies, also to babies born to HIV-positive mothers. BCG can cause disease (BCGosis) in HIV-infected babies. More importantly, BCG may also trigger immune responses in the body that lead to the spread of the HIV virus and early progression to AIDS.

Objective(s) and Hypothesis:

The researchers will investigate whether BCG causes progression of HIV by doing a clinical trial: babies born to HIV-positive mothers will be randomly allocated to get the BCG vaccine at birth or at 14 weeks of age. In these 2 groups of babies, the researchers will compare:

* The percentage of babies who progress to HIV disease
* Blood markers of HIV disease (the amount of virus and protective white blood cells in the body)
* The body's immune response to BCG vaccine and other childhood vaccines
* The percentage of children who develop BCG scarring, BCG vaccine complications and tuberculosis.

Potential Impact:

BCG is the most widely given vaccine worldwide and is routinely given to babies born to HIV-positive mothers in developing countries. Any effect that BCG has on HIV progression in babies will have a significant public health impact in settings with a high burden of HIV disease.

ELIGIBILITY:
Inclusion Criteria:

* Maternal HIV status verified
* Study consent
* Uncomplicated singleton pregnancy with delivery planned at local health facility
* Resident in study area

Exclusion Criteria:

* Active tuberculosis or tuberculosis contact in mother
* No consent
* Planning to move out of study area
* Not planning on delivering at local maternal obstetric unit
* Not planning on attending local baby clinic

Max Age: 48 Hours | Sex: All | Healthy Volunteers: No
Age Groups: Child
Enrollment: 180 (Estimated)
Dates: Start 2006-05; Primary Completion 2008-12 (Actual); Study Completion 2009-08 (Estimated)

PRIMARY OUTCOMES:
BCG-induced cellular immune responses | 1 year

SECONDARY OUTCOMES:
BCG scarring | 18 months
Serum antibody responses | 52 weeks
Tuberculosis incidence | 1 year

CONTACTS AND LOCATIONS:
Overall Officials: Anneke C Hesseling, MD, Principal Investigator — Desmond Tutu TB Centre, Dept. Pediatrics and Child Health, Stellenbosch University
Locations (1):
- Desmond Tutu TB Centre, Cape Town, Western Cape, South Africa